CLINICAL TRIAL: NCT00913822
Title: Bioavailability of Desipramine Hydrochloride Tablets
Brief Title: To Demonstrate the Relative Bioavailability of Desipramine Hydrochloride Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 870609D
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-06

CONDITIONS: Depression
Keywords: Antidepressant
MeSH Terms: conditions — Depression | interventions — Desipramine

ARMS (2):
- 1 (Experimental): Desipramine Hydrochloride 100 mg Tablets (Cord Laboratories)
  Interventions: Drug: Desipramine Hydrochloride 100 mg Tablets (Cord Laboratories)
- 2 (Active Comparator): Norpramin 100 mg Tablets (Merrell Dow Pharmaceuticals, Inc.)
  Interventions: Drug: Norpramin 100 mg Tablets (Merrell Dow Pharmaceuticals, Inc.)

INTERVENTIONS:
Drug: Desipramine Hydrochloride 100 mg Tablets (Cord Laboratories)
  Arms: 1
Drug: Norpramin 100 mg Tablets (Merrell Dow Pharmaceuticals, Inc.)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of Desipramine Hydrochloride tablets.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 1987-12; Primary Completion 1987-12 (Actual); Study Completion 1987-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Jules Kann, M.D., Principal Investigator — University of Pittsburgh